CLINICAL TRIAL: NCT07305987
Title: Phase III Clinical Study, to Evaluate the Efficacy and Safety of PRO-232 Ophthalmic Solution on the Ocular Surface of Patients Postoperative to Cataract Surgery by Phacoemulsification.
Brief Title: PRO-232 in Patients Subjected to Cataract Surgery
Acronym: PRO-232
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH232-1023/III
Record Dates: First submitted 2025-07-30; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cataract Extraction
MeSH Terms: interventions — Moxifloxacin; Vision, Ocular; dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: Phase III, parallel, controlled, comparative, double-blind, multicenter clinical study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-232 (Experimental): Two eyedroppers: one for PRO-232 and another for Placebo. Both will be administrated as follows: 1 drop four times a day (QID) with a minimum of four hours between applications, in the study eye for 14 days; with the exception of day 1 (the same day of the baseline visit), where a reduction in the interval between applications to a minimum of 3 hours per day will be allowed. A period of minimum 5 minutes between eyedropper administration will be required.
  Interventions: Drug: Moxifloxacin / Dexamethasone Ophthalmic Solution; Drug: Placebo
- Moxifloxacin / Dexamethasone (Active Comparator): Two eyedroppers: one for moxifloxacin and another for dexamethasone. Both will be administrated as follows: 1 drop four times a day (QID) with a minimum of four hours between applications, in the study eye for 14 days; with the exception of day 1 (the same day of the baseline visit), where a reduction in the interval between applications to a minimum of 3 hours per day will be allowed. A period of minimum 5 minutes between eyedropper administration will be required.
  Interventions: Drug: Moxifloxacin Hydrochloride, Ophthalmic; Drug: Dexamethasone phosphate

INTERVENTIONS:
Drug: Moxifloxacin / Dexamethasone Ophthalmic Solution — Moxifloxacin 0.5% / Dexamethasone phosphate 0.1% Ophthalmic solution
  Other Names: PRO-232
  Arms: PRO-232
Drug: Placebo — Same excipients as PRO-232, without active principles (moxifloxacin and dexamethasone)
  Arms: PRO-232
Drug: Moxifloxacin Hydrochloride, Ophthalmic — Moxifloxacin 0.5% Ophthalmic solution
  Arms: Moxifloxacin / Dexamethasone
Drug: Dexamethasone phosphate — Dexamethasone phosphate 0.1% Ophthalmic solution
  Arms: Moxifloxacin / Dexamethasone

SUMMARY:
The main objective of this study is to evaluate the efficacy and safety of the PRO-232 formulation manufactured by Laboratorios Sophia S.A. de C.V. on the ocular surface of postoperative cataract patients versus a concomitant administration of ophthalmic moxifloxacin and dexamethasone.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group, controlled clinical study designed to evaluate the efficacy and safety of PRO-232 ophthalmic solution in postoperative cataract patients. Participants will receive study treatment for 14 days.

The primary efficacy endpoint is to evaluate PRO-232 ophthalmic solution applied to the ocular surface of postoperative cataract patients, compared with concomitant administration of ophthalmic moxifloxacin and dexamethasone, by the proportion of patients with a grade 0 cellularity after 14 days of treatment.

Secondary outcomes include assessment of anterior chamber cellularity, ocular inflammation, eye pain using the Wong-Baker Faces® Visual Analog Scale, incidence of treatment-releated unexpected adverse events, best-corrected visual acuity (BCVA), and changes in intraocular pressure (IOP).

ELIGIBILITY:
Inclusion Criteria:

* To have the ability to voluntarily grant their signed informed consent (FCI).
* Being able and willing to comply with scheduled visits in the treatment plan and other study procedures.
* Being 18 years of age or older.
* Male or female.
* Women within childbearing age who do not have a history of bilateral tubaric obstruction, hysterectomy, or bilateral oophorectomy should ensure continued use (initiated ≥ 30 days prior to signing the ICF) of a hormonal contraceptive method or intrauterine device (IUD) during the study period.
* Having a postoperative diagnosis (unilateral, single eye) of cataract extraction by phacoemulsification with uncomplicated intraocular lens (IOL) placement** on the day prior to inclusion.
* Having an intraocular pressure ≥ 8 and ≤ 21 mmHg.

  * A complicated cataract surgery will be defined by study, as any procedure where the planned surgical technique has been modified or the use of vitrectomy has been required, an IOL has not been placed, a different IOL from the originally planned model has been placed or an IOL has been placed outside the capsular bag, remains of the lens have been left inside the eye, there was rupture of the posterior capsule with or without the presence of vitreous, or detachment of Descemet's membrane occured, there was disinsertion of the capsular pouch, or there was trauma to the iris or ciliary body during the surgical procedure. In the event of any other situation that could be considered a complication and that is not reflected in this list, the inclusion of said patient will be at the discretion of the researcher.

Exclusion Criteria:

* Allergy to any of the components of the investigational products or to any of the compounds used during testing.
* Surgery on both eyes during the same surgical period.
* Not having had surgery within a period of 24 hours before inclusion.
* Performing iridectomy, or injury to the pupillary sphincter during phacoemulsification surgery.
* History of use of eye drops between the end of surgery and the baseline visit.
* History of diagnosis of glaucoma or ocular hypertension.
* History of chronic or recurrent inflammatory eye disease (uveitis, iritis, iridocyclitis, etc.), eye inflammation or pain in the eye of study prior to surgery.
* Presence of corneal abrasion or ulceration.
* Use of topical or subconjunctival steroids or nonsteroidal anti-inflammatory drugs (NSAIDs), 24 hours prior to surgery and until the start of instillation of investigational medications.
* Use of steroids or systemic anti-inflammatory drugs within 14 days prior to surgery or if you plan to use them during the study period, or the presence of a diagnosis requiring the use of these medications during the study period.
* Use of blood thinners, systemic steroids, or immunomodulators within the past two weeks.
* Periocular injection of any steroid 4 weeks prior to initiation of investigational drug instillation or depot steroid use 2 months prior to initiation of investigational drug instillation.
* Presence or suspicion of viral, bacterial or fungal keratitis and/or conjunctivitis.
* Presence or suspicion of endophthalmitis.
* Presence or suspicion of anterior segment toxic syndrome.
* Severe corneal edema that does not allow the evaluation of the anterior chamber.
* Any disease or condition that requires the use of steroids by any route other than topical ophthalmic application.
* Patients with a single functional eye.
* Any condition or disease that, in the opinion of the main investigator, does not make the patient suitable for the study.
* Having participated in any investigational clinical study 30 days prior to inclusion in this study.
* Having previously participated in this same study.
* Having an active inflammatory or infectious disease at the time of study entry.
* Having unresolved eye injuries or trauma at the time of study entry.
* Use of antibacterial, antiviral, or antifungal agents by any route of administration within 30 days prior to study enrollment (including intracameral transsurgical antibiotics or administered to irrigation solution), or during the study.
* Use of pilocarpine and prostaglandin analogues.
* Secondary implantation or replacement of the intraocular lens (IOL) in the study eye.
* For women: being pregnant, breastfeeding, or planning to become pregnant within the study period.
* Be or have an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is employed by the research site or sponsor, and who is directly involved in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with grade 0 cellularity among interventions | Day 1, 3, 8 and 15.
  Using a slit lamp, a detailed assessment of cellularity in the anterior chamber of the eye will be performed. Using a 0.5 X 8.0mm beam of light directed obliquely the degree of cellularity will be measured. The grade of cellularity in the anterior chamber will be reported acording to the following scale: Grade Number of cells Grade 0 (≤ 5 cells), grade 1+ (5-10 cells [mild]), grade 2+ (11-20 [moderate]), grade 3+ (21-50 [marked]), grade 4+ (over 50 [severe]). The evaluated population for this outcome measure will be the PP population (subjects who finished the study without presenting any mayor deviations to protocol).
Proportion of patients presenting unexpected adverse events (AE) related between interventions | Day 1, 3, 8, 15 and 20.
  The manifested adverse events during the conduction of this trial will be obtained during trial visits and reported in the electronic CRF, where the clinical team of the center included the information from source documents. These will be previously checked by the monitor team, pharmacovigilance specialist, and the medical specialist part of the sponsor's crew to verify concordance with what was stipulated in the protocol. The classification as unexpected and/or related will be based in previously reported AE for the ingredients of the investigational products and comparators.
  This outcome measure considered the Intention-To-Treat (ITT) population, all participants who were randomized and exposed to treatment, regardless of whether they finished the study.

SECONDARY OUTCOMES:
Degree of cellularity in the anterior chamber between interventions | Day 1, 3, 8 and 15.
  Using a slit lamp, a detailed assessment of cellularity in the anterior chamber of the eye will be performed. Using a 0.5 X 8.0mm beam of light directed obliquely the degree of cellularity will be measured. The grade of cellularity in the anterior chamber will be reported acording to the following scale: Grade Number of cells Grade 0 (≤ 5 cells), grade 1+ (5-10 cells [mild]), grade 2+ (11-20 [moderate]), grade 3+ (21-50 [marked]), grade 4+ (over 50 [severe]). A higher score is a worse outcome.
  This outcome measure considered the Intention-To-Treat (ITT) population, all participants who were randomized and exposed to treatment, regardless of whether they finished the study.
Pain level score between interventions. | Day 1, 3, 8 and 15.
  The patient's level of eye pain will be assessed using a visual analog scale (Wong-Baker FACES® Visual Analog Scale). The scoring system will be as follows: Severity: (0) Doesn't hurt, (2) Hurts a little, (4) Hurts a little more, (6) Hurts a lot, (8) Hurts too much, (10) Unbearable pain. A higher score is a worse outcome.
  This outcome measure considered the Intention-To-Treat (ITT) population, all participants who were randomized and exposed to treatment, regardless of whether they finished the study.
Changes in best corrected visual acuity (BCVA) measurement between interventions | Day 1, 3, 8 and 15.
  The patient will be evaluated using his/her best refractive correction. BCVA is a test of visual function. It will be evaluated with the Snellen chart. The Snellen chart is the standard tool used to evaluate visual acuity. It was located in a place with adequate lighting, natural or artificial and at a distance of 3 meters from the subject to be evaluated. The contralateral eye to which it will be evaluated is covered, then the examiner detects until the line can clearly see the letters given he or she a score, the normal score for a VA is 20/20.This score can be expressed in fraction (i.e. 20/20) decimal (i.e. 1.0), or LogMAR (i.e. 0) formats. In this study, BCVA wiil be expressed in fraction and LogMAR formats. In fraction format and in LogMAR, a higher denominator number or number (respectively) is a worse outcome.
Proportion of patients who present an increase in intraocular pressure (IOP) ≥10 mmHg compared to baseline. | Day 1, 3, 8 and 15.
  The IOP will be measured through Goldmann tonometer in milligrams of mercury (mmHg). After instillation of topical anesthetic (tetracaine 0.5%) and fluorescein stain, IOP will be evaluated. Normal values are considered between 10 and 21 mmHg.

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Retina Center, Tijuana, Estado de Baja California
  - RGH Integra, Puebla City, Puebla

IPD SHARING:
Plan to Share IPD: No